CLINICAL TRIAL: NCT05952817
Title: The Effect of Virtual Reality on Pain, Physical Function, and Health-related Quality of Life in Children With Sickle Cell Disease: A Randomized Controlled Trial
Brief Title: Effect of Virtual Reality on Pain and Function in Children With Sickle Cell Disease: A Randomized Controlled Trial
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afnan Bkri (Other Government)
Responsible Party: Sponsor-Investigator, Afnan Bkri, Physiotherapist, Ministry of Health, Saudi Arabia
Organization: Ministry of Health, Saudi Arabia (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MohSaudiArabia1; Jazan health cluser ethics com (Other: R/N(H-10-Z-141))
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: SCD
Keywords: Sickle Cell Disease; Virtual Reality; Numeric Rating Scale; Randomized Controlled Trial; Children; Health-Related Quality of Life; Pain; Functional Mobility
MeSH Terms: conditions — Anemia, Sickle Cell; Pain

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned into two parallel groups following hospital discharge. The intervention group received a virtual reality (VR) program consisting of multiple sessions delivered over five weeks, while the control group continued with usual care. Both groups were followed at regular intervals, and outcome measures including pain intensity, physical function (Timed Up and Go), and health-related quality of life (PedsQL) were assessed at baseline, week 3, and week 5. The design followed a parallel assignment model without crossover between groups.
Who Masked: Outcomes Assessor
Masking Description: No additional parties were masked beyond the outcomes assessor. Only the assessor responsible for measuring clinical outcomes was blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- virtual reality treatment (Experimental): Participants assigned to this arm received a fully immersive virtual reality (VR) exercise program. The intervention consisted of a series of interactive physical therapy games designed to improve functional mobility, joint movement, balance, and pain management. Sessions were conducted at home over five weeks using an Oculus Quest 2 headset and KindVR Aqua software. Each session lasted 15 minutes and was supervised weekly by a pediatric physical therapist through follow-up communication.
  Interventions: Device: virtual reality
- Standard Care Group (No Intervention): Participants in this group received standard care without any additional VR-based interventions. They continued with their usual medical management and home routines as prescribed by their healthcare providers. No structured exercise or virtual therapy was provided during the study period.

INTERVENTIONS:
Device: virtual reality — Virtual reality (VR) technology is a new medical intervention technique founded on the principle of distraction, providing real perceptual stimuli such as visual images, spatial sounds, tactile, and sensory feedback stimuli.(Zhang et al., 2022)
  Arms: virtual reality treatment

SUMMARY:
Significance or rationale of the study:

Virtual reality (VR) is a promising non-pharmacological pain management tool. It enhances motor function by promoting cortical reorganization and neuroplasticity. Its multimodal biofeedback engages sensory and cognitive functions, making therapy interactive, motivating, and easy to understand. With strong rehabilitation potential, VR helps patients adapt to real-world movements (Laver, 2020). Initially used for procedural pain management, VR is now expanding into chronic pain rehabilitation by encouraging engagement with difficult or avoided movements (Griffin et al., 2020). Additionally, VR offers a dynamic alternative to traditional exercises, improving adherence and outcomes. Integrating entertainment into therapy can motivate children, enhancing their physical and psychological well-being. Recently, a few studies revealed an improvement in vaso-occlusive episodes (VOE) after VR treatment (Agrawal et al., 2019). However, efficacy studies are needed to assess VR's potential benefits. Additionally, data regarding VR's efficacy on daily pain, functional mobility, and HRQOL as complementary therapy are limited

DETAILED DESCRIPTION:
1. To investigate the effect of VR in reducing daily pain in children with SCD
2. To evaluate the impact of VR on improving functional mobility in children with SCD.
3. To examine the changes in PedsQL in children with SCD after engaging in VR experiences.
4. To evaluate the safety and satisfaction of fully immersive VR therapy in children with

ELIGIBILITY:
Inclusion Criteria:

1. Children aged between 8 and 13 years.
2. Diagnosed with sickle cell disease (SCD), including homozygous SCA and other clinically confirmed variants.
3. Medically stable and cleared by the treating physician to participate in mild activity.
4. Receiving hydroxyurea as part of routine care.
5. Able to follow simple instructions and communicate pain levels.
6. Parental/legal guardian consent and child assent obtained.

Exclusion Criteria:

1. Presentence of developmental, neurological, or genetic disorders.
2. History of hip replacement or major orthopedic conditions affecting mobility.
3. Current acute chest syndrome or unstable clinical condition.
4. Visual or hearing impairments that would interfere with VR use.
5. Participation in concurrent physiotherapy or rehabilitation programs.
6. Previously enrolled in phase one of the current study (if applicable)

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Pain Intensity (Numeric Rating Scale - NRS) | Baseline, Week 3, and Week 5
  Pain intensity was assessed using the validated Arabic version of the Numeric Rating Scale (NRS), which ranges from 0 (no pain) to 10 (worst imaginable pain). Participants were asked to rate their pain immediately before and after the VR session to measure the short-term analgesic effect of the intervention.

SECONDARY OUTCOMES:
Health-Related Quality of Life (PedsQL) | Baseline, Week 3, and Week 5
  The Pediatric Quality of Life Inventory (PedsQL) Generic Core Scale was used to assess health-related quality of life in children aged 8-13 years. The Arabic validated version was administered at baseline, mid-intervention (week 3), and post-intervention (week 5). Higher scores indicate better quality of life across physical, emotional, social, and school functioning domains.
Functional Mobility (Timed Up and Go Test - TUG) | Baseline, Week 3, and Week 5
  Functional mobility was measured using the Timed Up and Go (TUG) test. Participants were instructed to rise from a chair, walk 3 meters, turn around, walk back, and sit down. The total time taken to complete the task was recorded in seconds. Assessments were conducted at baseline, week 3, and week 5.

CONTACTS AND LOCATIONS:
Overall Officials: afaf Ah shaheen, PHD, Study Director — King Saud University
Locations (1):
- Prince Mohammed bin Nasser Hospital, Jizan, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD including pain scores and outcome measures will be available upon reasonable request with appropriate ethical approval.
  De-identified individual participant data (IPD), including pain scores and functional outcomes, will be made available upon reasonable request. Supporting documents such as the study protocol, statistical analysis plan, clinical study report, and analytic code will also be provided. Data will be shared through institutional data-sharing agreements and with approval from the responsible ethics committee. Availability is expected within 6 months following publication.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Individual participant data (IPD) and supporting documents will be made available beginning 6 months after publication of the main findings. Data will remain accessible for up to 3 years following the date of publication.
Access Criteria: Qualified researchers affiliated with academic institutions or healthcare organizations may request access to de-identified IPD and supporting documents (study protocol, SAP, CSR, and analytic code). Requests must include a data use agreement and be reviewed and approved by the institutional ethics committee. Approved data will be shared securely via institutional platforms or encrypted file transfer.

REFERENCES:
- [Background] Agrawal AK, Robertson S, Litwin L, Tringale E, Treadwell M, Hoppe C, Marsh A. Virtual reality as complementary pain therapy in hospitalized patients with sickle cell disease. Pediatr Blood Cancer. 2019 Feb;66(2):e27525. doi: 10.1002/pbc.27525. Epub 2018 Oct 26. PMID 30362236
- [Derived] Hassan AA, Algabbani MF, Farrag A, Elsayed W, Rezk MZA, Bindawas SM, Alhusaini AA, Shaheen AAM. Effect of fully immersive virtual reality on daily pain, functional mobility, and health-related quality of life in pediatric sickle cell disease: a single-blinded randomized clinical trial. Disabil Rehabil. 2026 Feb 10:1-15. doi: 10.1080/09638288.2026.2625551. Online ahead of print. PMID 41664928

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT05952817/Prot_SAP_000.pdf